CLINICAL TRIAL: NCT01908075
Title: REACH Fostair vs Seretide - Real-world Effectiveness of Combination Therapies in Primary Care Asthma Management
Brief Title: Real-world Effectiveness of Combination Therapies in Primary Care Asthma Management
Acronym: REACH
Status: Completed | Type: Observational
Sponsor: Research in Real-Life Ltd (Network)
Collaborators: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Principal Investigator, David Price, Prof., MD, Professor David Price, Research in Real-Life Ltd
Other Study IDs: R04312
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Last update posted 2013-07-25 (Estimated); Status verified 2013-07

CONDITIONS: Asthma
Keywords: Primary care; Asthma management; Real-world; Observational; Fostair; Seretide
MeSH Terms: conditions — Asthma | interventions — Fluticasone-Salmeterol Drug Combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- BDP/FOR: Patients receiving ICS/LABA therapy as FP/SAL (Seretide®) who, at an index prescription date (IPD): Change their therapy to BDP/FOR (Fostair®) at same or lower BDP-equivalent ICS dose
  Interventions: Drug: FP/SAL; Drug: BDP/FOR
- FP/SAL: Patients receiving ICS/LABA therapy as FP/SAL (Seretide®) who, at an index prescription date (IPD) : Remain on FP/SAL at the same BDP-equivalent ICS dose
  Interventions: Drug: FP/SAL

INTERVENTIONS:
Drug: FP/SAL
  Other Names: Seretide®
Drug: BDP/FOR
  Other Names: Fostair® 100/6
  Groups: BDP/FOR

SUMMARY:
To evaluate whether beclomethasone dipropionate / formoterol (BDP/FOR; Fostair® 100/6) is at least equivalent in terms of exacerbation prevention to fluticasone dipropionate / salmeterol (FP/SAL; Seretide® 125) in matched asthma patients switching to BDP/FOR following treatment with FP/SAL in normal clinical practice compared with patients not switched.

DETAILED DESCRIPTION:
To evaluate whether beclomethasone dipropionate / formoterol (BDP/FOR; Fostair® 100/6) is at least equivalent in terms of exacerbation prevention to fluticasone dipropionate / salmeterol (FP/SAL; Seretide®) in matched asthma patients switching to BDP/FOR following treatment with FP/SAL in normal clinical practice compared with patients not switched. To evaluate respiratory outcomes for Fostair in comparison to Seretide using a UK primary care database (in patients switched for cost rather than clinical reasons).

ELIGIBILITY:
Inclusion Criteria:

* Aged: 18-80 years 61-80 years to be non-smokers only
* Evidence of asthma: a diagnostic code for asthma or two scripts for asthma..
* Baseline FP/SAL therapy: ≥2 prescription for ICS/LABA therapy as FP/SAL
* Evidence of Continuing Therapy: Include only patients who receive ≥2 prescriptions for the therapy under study during the outcome year (i.e. ≥1 prescription at the index date and ≥1 other). UK average is 3-4 prescriptions refilled per year, so ≥2 ensures capture of "real-life" data.
* Evidence of Switching for economic reasons: FP/SAL patients from practices with ≥5 switches to Fostair in a 3 month period to minimise data taken from switching of anomalous patients; optimal practices for inclusion are those switching "wholesale" for economic reasons.

Exclusion Criteria:

* Any chronic respiratory disease other than asthma
* Are receiving maintenance oral steroid therapy during baseline period

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients are diagnosed with asthma or COPD and aged between 18-80 years with all 61-80 year olds being non-smokers only
Sampling Method: Non-Probability Sample
Enrollment: 194723 (Actual)
Dates: Start 2011-01; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Exacerbations : rate ratio | 1 year
  Where an exacerbation is defined as:
  (i) Asthma-related
  1. Hospital attendance / admissions OR
  2. Accident & Emergency (A&E) attendance OR (ii) Use of acute oral steroids.
  Where:
  * ≥1 oral steroid prescription occurs within 2 weeks of another, or
  * ≥1 hospitalisation occurs within 2 weeks of another, or
  * ≥1 hospitalisation occurs within 2 weeks of an oral steroid prescription

SECONDARY OUTCOMES:
Exacerbation control | 1 year
  Proxy Asthma Control. The absence of exacerbation and the absence of antibiotic prescribing for lower respiratory tract infections (often a pragmatic prescribing decision taken by GPs in real world practice).
  Controlled:
  (i) No Asthma-related:
  1. Hospital attendance or admission
  2. A&E attendance, OR
  3. Out of hours attendance, OR
  4. Out-patient department attendance (ii) GP consultations for lower respiratory tract infection (iii) Prescriptions for acute courses of oral steroids
  Uncontrolled:
  (i) All others.
  a. Proxy Asthma Control + SABA As above, but with an additional criterion that limits "controlled" patients to those who use ≤200mcg salbutamol daily.
Proxy asthma control + SABA | 1 year
  As above, but with an additional criterion that limits "controlled" patients to those who use ≤200mcg salbutamol daily
Treatment success | 1 year
  No exacerbation and no change in therapy during the outcome year, where changes are:
  •≥50% increase in ICS dose relative to IPD dose, and/or
  * Change in ICS/LABA drug within class, and/or
  * Change in delivery device, and/or
  * Use of additional (defined as not received during baseline year) therapy as defined by: theophylline, leukotriene receptor antagonists (LTRAs).
Asthma Control (including SABA) | 1 year
  Defined as proxy asthma control (above) plus:
  Average daily prescribed dose of ≤200mcg salubtamol / ≤500mcg terbutaline
Hospitalisations | 1 year
  Asthma-related hospitalizations
  * Definite: Hospitalisations coded with an asthma read code
  * Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of an asthma read code
  Respiratory hospitalisations
  * Definite: Hospitalisations coded with a lower respiratory code relevant for Paeds (for example J450)
  * Definite + Probable: Hospitalisations with an asthma read code + uncoded hospitalisations occurring within a 7-day window (either side of the hospitalisation date) of a lower respiratory read code
Medication possession ratio | 1 year
  For ICS, defined as the number of days supply of ICS / 365 x 100%
  Controller/reliever ratio: number of controller units/ number of controller units + number of reliever units. Controllers are defined as ICS (including fixed combination ICS/LABA) and LTRA, while relievers are SABA. For ICS a unit is taken to be one inhaler; for LTRA a unit is one prescription.

CONTACTS AND LOCATIONS:
Overall Officials: David Price, Principal Investigator — University of Aberdeen